CLINICAL TRIAL: NCT06443593
Title: Vitamin B12, Vitamin D and Iron Supplementation for Improvement of Nerve Conduction Velocities in Children and Youth With Type 1 Diabetes
Brief Title: Effect of Micronutrient Supplementation on Nerve Conduction Velocity in T1D- RCT
Acronym: NCVRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, Consultant Pediatrician and Deputy Director, Hirabai Cowasji Jehangir Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JCDC/BHR/24/014
Record Dates: First submitted 2024-05-16; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
Keywords: Diabetic neuropathy; children and youth with type 1 diabetes; vitamin B12; vitamin D; oral iron; Nerve conduction velocity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Only vitamin B12 supplements (Active Comparator): Only vitamin B12 supplements 2.2 mcg OD for 24 weeks
  Interventions: Dietary Supplement: Tablet VitaBliss vitamin B12 (2.2 mcg)
- Arm 2: Vitamin B12 and oral iron supplements (Active Comparator): Vitamin B12 2.2 mcg OD daily and oral iron 25 mg OD daily for 24 weeks
  Interventions: Dietary Supplement: Tablet VitaBliss vitamin B12 (2.2 mcg) and Syrup Orofer (5 ml = 50 mg)
- Arm 3: Vitamin B12 and vitamin D3 (Active Comparator): Vitamin B12 2.2 mcg OD daily and vit D3 60,000 IU once in three months for 24 weeks
  Interventions: Dietary Supplement: Tablet VitaBliss vitamin B12 (2.2 mcg) and Tablet Tayo (60000 IU)

INTERVENTIONS:
Dietary Supplement: Tablet VitaBliss vitamin B12 (2.2 mcg) — Oral vitamin B12 supplement 2.2 mcg from BLISS WELNESS, Bliss Lifesciences, LLP to be administered once daily for 24 weeks
  Arms: Arm 1: Only vitamin B12 supplements
Dietary Supplement: Tablet VitaBliss vitamin B12 (2.2 mcg) and Syrup Orofer (5 ml = 50 mg) — Oral vitamin B12 supplement 2.2 mcg from BLISS WELNESS, Bliss Lifesciences, LLP to be administered once daily for 24 weeks and oral iron 25 mg from Emcure Pharmaceuticals Ltd. to be administered once daily for 24 weeks
  Arms: Arm 2: Vitamin B12 and oral iron supplements
Dietary Supplement: Tablet VitaBliss vitamin B12 (2.2 mcg) and Tablet Tayo (60000 IU) — Oral vitamin B12 supplement 2.2 mcg from BLISS WELNESS, Bliss Lifesciences, LLP to be administered once daily for 24 weeks and oral vitamin D3 (60000 IU) from Eris Lifesciences Ltd to be administered once in 3 months for 24 weeks
  Arms: Arm 3: Vitamin B12 and vitamin D3

SUMMARY:
Type 1 diabetes can complicate to peripheral neuropathy due to preferential involvement of small unmyelinated nerve fibers (pain and temperature sensation) followed by myelinated nerve fibers (vibration and proprioception). The SEARCH for diabetes in youth study found diabetic neuropathy in 7% of T1D youth. The clinical form of peripheral neuropathy is rare in childhood and pathophysiological changes begin during childhood and accelerate in puberty. Adolescents with these changes can be picked up more reliably by electrophysiological studies than by clinical examination. Nerve conduction studies are the gold standard diagnostic tests for detection of peripheral neuropathy. Role of vitamin B12 in nerve regeneration is well known while causal association of vitamin D deficiency in type 1 diabetes and its role in axonal degeneration is also reported. The previous ongoing studies from authors' group have shown relationship between poor oral iron intake and subclinical neuropathy in children with type 1 diabetes (manuscript in submission). The present randomised clinical trial is aimed at assessing vitamin B12, vitamin D and iron supplementation for improvement of nerve conduction velocities in children and youth with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Children/ parents/ youth willing to participate in the study with an informed consent/ assent.
2. Children/ youth Age > 10 years
3. Diabetes duration > 2 years
4. Diagnosed with type 1 diabetes

Exclusion Criteria:

1. Age < 10 years
2. Diabetes duration < 2 years
3. Children/ youth receiving vitamin B12, vitamin D and/or oral iron supplements
4. Children/ youth with any other disease condition involving nerve or muscle function
5. Children/ parents/ youth not willing to consent to participate in the study.

Ages: 10 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-02-08 (Estimated); Study Completion 2025-02-08 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction velocity | 6 months
  Change in nerve conduction velocity of children and adolescents with type 1 diabetes after supplementation with vitamin B12, oral iron and vitamin D
Serum vitamin B12, serum ferritin, serum vitamin D3 | 6 months
  Change in serum vitamin B12, serum ferritin, serum vitamin D3 levels using standardized assays in children and adolescents with type 1 diabetes after supplementation with vitamin B12, oral iron and vitamin D

SECONDARY OUTCOMES:
Dynamic muscle function | 6 months
  Maximum relative power (watt/kg) will be assessed using jumping mechanography
Dynamic muscle function | 6 months
  Maximum relative force (Newton/kg) will be assessed using jumping mechanography
Glycemic control (HbA1c) | 6 months
  Glycemic control will be assessed using glycated hemoglobin (HbA1c) by standardized assays

CONTACTS AND LOCATIONS:
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No